CLINICAL TRIAL: NCT05911542
Title: Dentists' Attitudes Towards Pharmacological Management of Acute Pain in Children and Adolescents - a Follow-up Survey
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Sponsor
Other Study IDs: FO 2021/536
Record Dates: First submitted 2023-06-07; First posted 2023-06-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Dental Practitioners: Participants are asked to complete a survey about pain management strategies.
  Interventions: Behavioral: Survey
- Specialist Paediatric Dentists: Participants are asked to complete a survey about pain management strategies.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Participants complete survey about pain management practices

SUMMARY:
The aim of this study is to investigate Swedish dentists' attitudes about pain management when treating children and adolescents by assessing 1) dentists' recommendations for the use of pre- and postoperative analgesics, (2) use of local anaesthesia during treatment of primary and permanent teeth, and (3) if the use of these strategies differs between General Dental Practitioners (GDP) and Specialist Paediatric Dentists (SPD).

All Swedish SPDs (including post-graduate dentists in paediatric dentistry), circa 150 in total, and approximately 1,000 GDPs in County Skåne, Sweden will be invited to answer a questionnaire.

DETAILED DESCRIPTION:
This survey study is follow-up to a survey carried out in 2014, addressed to Swedish General Dental Practitioners (GDPs) and Specialist Paediatric Dentists (SPDs). The aim of this study is to investigate Swedish dentists' attitudes about pain management when treating children and adolescents by assessing 1) dentists' recommendations for the use of pre- and postoperative analgesics, 2) use of local anaesthesia during treatment of primary and permanent teeth, and 3) if the use of these strategies differs between GDPs and SPDs.

All SPDs (including post-graduate dentists in paediatric dentistry) in Sweden, circa 150 in total, and approximately 1,000 GDPs, will be invited to answer the questionnaire. To be included GDPs need to have registered addresses in county Skåne, Sweden, and be accredited to provide dental care to children and adolescents by Region Skåne, the regional public health and dental care provider. A questionnaire along with written information about the study and two consent forms will be mailed to presumptive study participants. Those willing to participate in the study are asked to return (postage prepaid) one signed consent form and the completed questionnaire. The questionnaire is adapted from one previously used in Sweden. It contains demographic questions, and questions regarding work situation. These questions are followed by four clinical scenarios, and questions relating to use of pain management practices. Responses are given on a 5-point Likert scale. The final questions are open ended and concern the use of pre- and postoperative analgesics.

ELIGIBILITY:
Inclusion Criteria:

General Dental Practitioners with a civil registration address in County Skåne, Sweden.

Specialist Paediatric Dentists in Sweden.

Exclusion Criteria:

Not accredited to provide dental care to children and adolescents (applies to General Dental Practitioners).

≥ 65 years of age

Max Age: 64 Years | Sex: All
Age Groups: Child, Adult
Study Population: General Dental Practitioners with a civil registration address in County Skåne, Sweden, and Specialist Paediatric Dentists in Sweden.
Sampling Method: Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Attitudes towards management of acute pain | 4 months
  Dentists' attitudes towards pharmacological management of acute pain in children and adolescents measured on a 5 point Likert scale, ranging from 'always' to 'never'.

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Klingberg, Professor, Principal Investigator — Malmö University
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berlin H, List T, Ridell K, Klingberg G. Dentists' attitudes towards acute pharmacological pain management in children and adolescents. Int J Paediatr Dent. 2018 Mar;28(2):152-160. doi: 10.1111/ipd.12316. Epub 2017 Jul 10. PMID 28691744
- [Background] Wondimu B, Dahllof G. Attitudes of Swedish dentists to pain and pain management during dental treatment of children and adolescents. Eur J Paediatr Dent. 2005 Jun;6(2):66-72. PMID 16004534